CLINICAL TRIAL: NCT00925912
Title: A Randomized Clinical Trial of Closed Hemorrhoidectomy Under Local Perianal Block Versus Spinal Anesthesia
Brief Title: A Trial of Closed Hemorrhoidectomy Under Local Perianal Block Versus Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: s023h/49
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Postoperative Pain; Complications; Satisfaction
Keywords: Hemorrhoidectomy; perianal block; local anesthesia; spinal anesthesia
MeSH Terms: conditions — Pain, Postoperative; Personal Satisfaction | interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): spinal anesthesia: Active Comparator
  The SA group were received a subarachnoid block with 1.5-2.0 ml of 0.5% bupivacaine.
  Interventions: Procedure: spinal block
- 2 (Experimental): Perianal block with 0.25% bupivacaine
  Interventions: Procedure: Perianal block

INTERVENTIONS:
Procedure: spinal block — 0.5% bupivacaine 1.5-2 ml injected to subarachnoidal space
  Other Names: marcaine 0.5%
  Arms: 1
Procedure: Perianal block — 0.25% bupivacaine injected at perianal region
  Other Names: Marcaine 0.25%
  Arms: 2

SUMMARY:
Hemorrhoidectomy can be carried out under several modes of anesthesia. In western country hemorrhoidectomy usually be performed under general anesthesia, however there may be the complications resulted from general anesthesia together with associated diseases in advanced age, caudal or spinal anesthesia has been used as an alternative to general anesthesia (GA) for hemorrhoid surgery but they all require a trained anesthetist and have numerous known complications. Since, anesthesiologists are not always available then local anesthesia is an alternative mode of anesthesia that surgeon can safely carry out by their own. Local anesthetic produce a loss of sensation and muscle paralysis in a circumscribed area of body by localized effect on peripheral nerve endings. The local anesthesia is able to provide fully relaxation of the anal canal which is an ideal setting for various anal surgical procedures. The results of hemorrhoid surgery under this mode of anesthesia have been demonstrated in many publications. Local anesthesia is a safe and effective technique while fewer risks and complications compared with general or spinal anesthesia. In Thailand both spinal anesthesia and local perianal block have routinely been used for various kinds of anorectal surgery. However, so far there has no any trial conducting to compare between these two techniques.

DETAILED DESCRIPTION:
Objectives: To study analgesic efficacy, postoperative voiding problems, patients' satisfaction, and other complications after closed hemorrhoidectomy comparison between local perianal block and spinal anesthesia.

Research design: Randomized controlled trial Setting: Phramongkutklao Hospital Research methodology: A total of 64 subjects (32 males and 32 females) underwent elective hemorrhoidectomy were randomly allocated into two groups. Thirty-two patients were randomly allocated to receive spinal anesthesia (SA group) while 32 patients received local perianal block (LA group). Duration of analgesic effect, pain measurement with visual analogue scale (VAS) at 6 and 24 hours, quantity of analgesic medication administered, postoperative complication, and patient's satisfaction with the anesthetic technique were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 60 years with grade 3 or 4 hemorrhoid.
2. Had no history of bupivacaine allergy.

Exclusion Criteria:

1. Complicated hemorrhoid e.g. prolapsed or incarcerated hemorrhoid, gangrenous hemorrhoid.
2. Associated anorectal disease.
3. Patients whose characteristics of his/her buttock were difficult to gained adequate exposure when performing surgery under local anesthesia such as the mounds of his/her buttock is very high and rise almost straight up from the anal verge.
4. Patient was unfit for surgery e.g. heart disease, liver cirrhosis, or coagulopathy.
5. Patients who had symptoms of benign prostatic hypertrophy or bladder neck obstruction.
6. Pregnancy.
7. Patients with neuropsychotic problems.
8. Did not agree to participate this study

Ages: 18 Years to 60 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2006-12; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The degree of pain measured by visual analogue scale at 6 and 24 hrs after surgery. | within 24 hrs

SECONDARY OUTCOMES:
Patients' satisfaction with the anesthetic techniques, postoperative voiding complications, and other complications | within 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Sahaphol Anannamcharoen, M.D.,M.Sc., Principal Investigator — Phramongkutklao College of Medicine and Hospital